CLINICAL TRIAL: NCT01998529
Title: A Phase I Study of Cytoreductive Surgery and Hyperthermic Intrathoracic Pleural Chemotherapy (HITC) With Escalating Doses for Children and Adolescents With Unilateral Pleural Malignancy
Brief Title: Study of Cytoreductive Surgery and Hyperthermic Intrathoracic Pleural Chemotherapy (HITC) With Escalating Doses for Children and Adolescents With Unilateral Pleural Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0657; NCI-2014-00510 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-11-19; First posted 2013-11-29 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Unilateral Pleural Malignancy; Metastatic active pleural malignancy; Lung tumors; Sarcomas; Cytoreductive Surgery; Hyperthermic Intrathoracic Pleural Chemotherapy; HITC; Cisplatin; Platinol-AQ; Platinol; CDDP; Amifostine; Ethyol; Ethiofos; Gammaphos
MeSH Terms: conditions — Lung Neoplasms; Sarcoma | interventions — Cisplatin; Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cisplatin (Experimental): After cytoreductive surgery, possible pneumonectomy, and possible diaphragm resection, the chest cavity will be closed in layers, leaving inflow and outflow chest tubes in place. Catheters connected to an extracorporeal perfusion circuit. Starting dose of hyperthermic cisplatin 120 mg/m2. Perfusion continued for 60 minutes after adding the cisplatin at a target temperature of 41 C (+0.5 C). In order to limit the systemic toxicity of cisplatin, amifostine administered intravenously over 15 minutes beginning 30 minutes after cisplatin perfusion. Patient response to amifostine continuously monitored by anesthesiologist. Infusion may be stopped and/or restarted based on blood pressure.
  Interventions: Drug: Cisplatin; Drug: Amifostine

INTERVENTIONS:
Drug: Cisplatin — Starting dose of hyperthermic cisplatin 120 mg/m2. Perfusion continued for 60 minutes after adding the cisplatin at a target temperature of 41 C (+0.5 C).
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Amifostine — Amifostine administered intravenously over 15 minutes beginning 30 minutes (+ 15 minutes) after the cisplatin perfusion.
  Other Names: Ethyol; Ethiofos; Gammaphos

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of heated cisplatin that can be given to patients with lung tumors. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Surgery and Study Drug Administration:

If you are found to be eligible to take part in this study, chest surgery will be performed to try to remove as many tumors as possible. The chest surgery is not being performed specifically for this research study and would be performed as part of your standard of care treatment even if you didn't take part in this study. You will be given a separate consent form to sign that explains the details and risks of chest surgery in more detail.

During the chest surgery, you will receive amifostine by vein to help prevent possible side effects, such as ear and/or kidney damage. The chest will then be closed with a plastic tube left in place. Then, the chest wash will begin. During the chest wash, a pump that is connected to the plastic tube pushes the heated cisplatin into the chest and then pulls it out to recirculate the cisplatin. The surgeon will also wash over the closed area of the surgical site with heated cisplatin. The heated cisplatin will be recirculated in and out of the chest over 60 minutes while the surgeon gently presses on the chest wall to help the cisplatin reach all areas in the chest. The plastic tube the heated cisplatin will be pumped through will stay in place after the surgery to drain the extra fluid. These are the same plastic tubes that would be present even if you did not agree to take part in this study.

During the surgery, extra blood (about ½ teaspoon each time) and fluid from the chest area will be collected for pharmacokinetic (PK) testing when you begin to receive the first infusion of the heated cisplatin, then 30 and 60 minutes after the infusion has started, and again 24 hours after receiving the heated cisplatin. The blood and fluid from the chest area will be collected through already placed catheters, so no additional needle sticks will be required. PK testing measures the amount of study drug in the body at different time points.

There is a chance that the surgeon may decide during the surgery that the chest wash will not be performed, for example if the disease has spread to or attached to certain organs. If this occurs, your doctor will discuss other treatment options with you after the surgery is complete.

Study Visits:

On Days 1-5, 11, and 14, (Day 1 being the day after surgery):

* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have a physical exam.

Follow-Up Visits:

About 1 month after the surgery is complete, you will have a follow-up visit and the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 1-3 teaspoons) will be drawn for routine tests.
* You will have a hearing test at the 1 month visit only.

It is recommended that you have follow-up visits at MD Anderson at 3 and 6 months after surgery. In addition to blood draws (about 1-3 teaspoons), you will have an MRI, CT, or PET-CT scan to check the status of the disease. These 3 and 6 month visits after surgery may be performed at your local doctor's office and/or laboratory.

Length of Study:

You will remain on study for up to 6 months. You will be taken off study if the disease gets worse.

If the study doctor learns that the disease has come back or gotten worse at the 6 month follow-up visit, you may be eligible to have the operation with heated cisplatin wash repeated. If you are eligible for to have the surgery repeated, your active participation on this study will end and then you will be given a new consent form to sign in order to be re-enrolled back onto this study.

This is an investigational study. Cisplatin is FDA-approved and commercially available for the treatment of advanced bladder cancer, metastatic testicular cancer, metastatic ovarian cancer, hepatoblastoma, neuroblastoma, metastatic appendiceal cancer, and abdominal mesothelioma. The use of a heated cisplatin wash during chest surgery in patients with lung tumors is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 3 years to </= 21 years.
2. Histologically or genetically proven unilateral primary or metastatic active pleural malignancy.
3. Radiologic workup must demonstrate that the thoracic disease is confined to only one hemi-thoracic cavity and must be deemed potentially resectable by the surgical team.
4. The extrathoracic disease must be controlled.
5. Patients must have a minimum expected duration of survival of 8 weeks as determined and documented by the attending surgeon or medical oncologist.
6. Patients must not have any systemic illness which precludes them from being an operative candidate.
7. Patients must have Adequate Renal Function Defined as: Creatinine clearance or radioisotope GFR >/=70ml/min/1.73 m^2 or a serum creatinine based on age/gender less than listed value in the table below: 1 to < 2 years 0.6 mg/dL for both males and females, 2 to < 6 years 0.8 mg/dL for both males and females, 6 to < 10 years 1 mg/dL for both males and females, 10 to < 13 years 1.2 mg/dL for both males and females, 13 to < 16 years 1.5 mg/dL for males and 1.4 mg/dL for females, >/= 16 years 1.7 for males and 1.4 for females
8. Patients will be eligible if the WBC is >/=1500/µl or ANC is >/=1,000 and platelets are >/= 50,000/mm^3
9. Adequate Liver Function Defined as: -Bilirubin (sum of conjugated + unconjugated) </= 1.5 x upper limit of normal (ULN) for age -SGPT (ALT) </=110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L. -Serum albumin >/= 2 g/dL.
10. Patients must be recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy and be at least 14 days past the date of their last treatment

Exclusion Criteria:

1. Patients will be ineligible if they have any concomitant cardiopulmonary disease which would place them at unacceptable risk for a major surgical procedure
2. Patients who have failed previous hemi-thoracic platinum therapy will be ineligible ("Failed" is having disease recurrence </= 3 months).
3. No pregnant or lactating females.
4. Patients will be ineligible if they have a lymphoma diagnosis.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Hyperthermic Intrathoracic Pleural Chemotherapy (HITC) | Change in dose levels at 30 and 60 minutes after the infusion has started, and again 24 hours after receiving the heated cisplatin
  If 2 dose limiting toxicities (DLTs) are observed at a given dose level, MTD has been exceeded. Dose level below expanded to a total of 6 patients and if </= 1 out of 6 patients experience a DLT at this dose level, this will be defined as the MTD.
  Dose limiting toxicity may occur at any time during the initial hospitalization before discharge following the HITC. The dose limiting toxicity is defined two ways. Hematologic DLT is defined as Grade IV neutropenia, anemia, or thrombocytopenia. Non-hematologic DLT is any Grade III or IV non-hematologic toxicity excluding Grade III nausea or vomiting, Grade III hepatic toxicity which returns to Grade I within four weeks of the HITC, or before hospital discharge, or Grade III fever occurring after the HITC.

SECONDARY OUTCOMES:
Time to Relapse | 3 months
  Evaluation of measurable disease performed 3 months and 6 months postoperatively (+2 weeks) using CT and physical exam. Disease progression defined by radiographically visible nodules greater than 1.5 cm.

CONTACTS AND LOCATIONS:
Overall Officials: David Rice, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org